CLINICAL TRIAL: NCT00080392
Title: Modulation of Vascular Endothelial Growth Factor (VEGF) Using an Engineered Zinc-Finger Transcription Factor to Treat Lower Limb Intermittent Claudication
Brief Title: EW-A-401 to Treat Intermittent Claudication
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040143; 04-H-0143
Record Dates: First submitted 2004-03-30; First posted 2004-03-30 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2011-12-29

CONDITIONS: Intermittent Claudication; Arteriosclerosis
Keywords: Gene Transfer; Therapeutic Angiogenesis; Peripheral Arterial Disease; Perfusion; Magnetic Resonance Imaging; Peripheral Vascular Disease; Claudication; PAD; Leg Claudication; Intermittent Claudication
MeSH Terms: conditions — Intermittent Claudication; Arteriosclerosis; Peripheral Arterial Disease; Peripheral Vascular Diseases

INTERVENTIONS:
Drug: DNA Plasmid Vector
Drug: EW-A-401 DNA Plasmid Vector

SUMMARY:
This study will test the safety of a drug called EW-A-401 in patients with intermittent claudication - pain and discomfort in the legs due to blockages of the arteries. The study will also evaluate whether EW-A-401 improves blood flow to the legs. EW-A-401 contains genetic material (DNA) that instructs the body to produce specific proteins that promote the growth of new blood vessels and may, therefore, improve blood flow to the legs.

Patients 21 years of age and older with pain or discomfort of one or both legs due to blockages of the arteries below the groin may be eligible for this study. Candidates are screened with a medical history, physical examination, blood and urine tests, eye examination, chest x-ray and CT scan of the chest, and treadmill tests. Patients who are able to exercise more than 12 minutes on the treadmill may not enroll in the study.

Participants undergo the following procedures:

* Muscle biopsy: On the first day of the study, patients have a muscle biopsy. This procedure is done under local anesthesia with mild sedation. A 1-inch incision is cut into the skin over a calf muscle and a small amount of muscle tissue is removed for examination by a pathologist.
* Drug treatment and tests: About 10 to 13 days after the biopsy, patients are admitted to the NIH Clinical Center for 3 to 5 days for drug treatment and tests. They receive 10 injections of either the study drug (EW-A-401) or placebo (an inactive substance) in each leg during a single session lasting about 1 hour. In addition, they have blood and urine tests, complete questionnaires about their symptoms, and undergo magnetic resonance imaging (MRI), a test that a magnetic field and radio waves to produce detailed images of body tissues and organs. For this procedure, the patient lies on a table that slides into the scanner (a large hollow tube) for imaging of the blood vessels in the legs. Patients wear headphones to muffle loud knocking and thumping sounds that occur during the scanning process.
* 30-day follow-up: Patients return to the Clinical Center three times over 30 days following the hospital stay for a medical history, physical examination, and blood and urine tests to assess the safety of EW-A-401.
* Extended follow-up: Patients return to the Clinical Center at 3, 6, and 12 months after hospitalization for a medical history and physical examination, blood and urine tests, two treadmill tests, questionnaires about symptoms, and MRI studies, including imaging for blood flow measurement. Blood flow to the legs is measured during MRI using large blood pressure cuffs inflated around the legs during the scanning. The cuffs are inflated very tightly for 5 minutes, and then a dye is injected into an arm vein to brighten the images. Additional pictures are taken over the next 5 to 10 minutes. At two of these follow-up visits, patients also have an eye examination, and at the 3- or 6-month visit they have a repeat muscle biopsy of the calf.

The study lasts 12 months. After 6 months, patients will be told whether they received EW-A-401 or placebo. Because EW-A-401 is so new, patients will continue to be contacted every year after the study is completed.

DETAILED DESCRIPTION:
Lower limb intermittent claudication, muscular pain with exercise relieved promptly by rest, is a disabling syndrome affecting over 10 million patients in the United States. Intermittent claudication is caused by peripheral artery atherosclerosis, the same disease causing heart attack. Peripheral artery atherosclerosis impairs blood flow to skeletal muscles in the lower limbs. Growth factors, such as vascular endothelial growth factor (VEGF-A), have been shown in animal studies to improve blood flow the lower limbs by promoting the growth of new blood vessels.

This clinical study tests the safety and feasibility of gene transfer of an agent (EW-A-401) intended to improve blood flow in the skeletal muscle of subjects with intermittent claudication. The investigational agent is a circle of genetic material (plasmid DNA) that instructs the body to produce a genetically-engineered transcription factor, a protein that regulates expression of genes. This specific transcription factor has been shown in animal studies to increase expression of the VEGF-A gene, and to promote the growth of new blood vessels. The study agent will be delivered by injection into leg muscle during a single session. This is the first human experience using this transcription factor.

This study has a randomized, double-blind, dose-escalation, placebo-controlled design. The primary outcome measure will be safety and toxicity. In addition, we will collect exploratory effectiveness information including blood flow, walking capacity, quality of life, and inspection of blood vessels on samples of leg muscle.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Adults greater than or equal to 21 years.
  2. Limiting lower limb intermittent claudication due to infra-inguinal obstructive atherosclerosis, not optimal for catheter-based treatment.
  3. Patient femoral artery inflow by radio contrast or magnetic resonance angiography within the previous 12 months.
  4. Stable symptoms for at least 4 months.
  5. Peak walking time (PWT) on standardized Gardner Exercise Treadmill Exam between 1 and 12 minutes.
  6. Resting ankle-brachial systolic blood pressure index (ABI) less than 0.9 in the more-affected limb.
  7. Bilateral PAD for subjects enrolled into Strata C-F with the less-affected limb having any of the following:
* Resting or post-exercise ABI less than or equal to 0.9.
* Typical intermittent claudication.
* Infrainguinal obstructive atherosclerosis in a femoropopliteal and/or tibial artery greater than or equal to 70%.

Subjects enrolled into Strata A and B may have both unilateral or bilateral peripheral atherosclerotic disease.

EXCLUSION CRITERIA:

1. Any history of malignancy or a known genetic predisposition for developing cancer except for curatively resected basal cell carcinoma of skin, squamous cell carcinoma of skin, cervical carcinoma in situ, or resected benign colonic polyps.
2. Non-compressible arteries (resting ankle-brachial systolic blood pressure index (ABI) greater than 1.3 in the more-affected limb).
3. Evidence of malignancy after screening according to modified American Cancer Society Guidelines in the following organ systems (screening procedures in addition to history and physical exam are noted):

   -Prostate: subjects with the following PSA levels above the recommended age-specific cut-points will be excluded

   Age 50-59 greater than or equal to 3.7

   Age 60-69 greater than or equal to 5.1

   Age 70-79 greater than or equal to 7.0

   Age 80 plus-greater than or equal to 7.2

   Subjects with PSA values above the age-specific cut-points are eligible if a prostate biopsy, within 12 months, shows neither prostate cancer nor high-grade prostatic intraepithelial neoplasia (PIN).
   * Breast: mammogram
   * Cervix: Pap smear
   * Colon: Colonoscopy
   * Skin
   * Lung: contrast chest CT scan
4. Proliferative retinopathy, severe non-proliferative retinopathy, advanced age-related macular degeneration, especially subjects with chorodial neovascularization, diabetic retinopathy, macular edema, or intraocular surgery within 3 months.
5. Limiting symptom on Gardner Exercise Treadmill Examination other than intermittent claudication.
6. Co-morbid conditions that limit exercise capacity:

   * Severe arthritis affecting lower extremities
   * Severe chronic obstructive pulmonary disease
   * Angina pectoris greater than Canadian Angina Class 2
   * Dyspnea greater than New York Heart Association Class II
7. Cardiovascular surgery or percutaneous revascularization within 4 months.

   * Inclusion is permitted two or more months after successful iliac stenting in the presence of significant infra-inguinal atherosclerotic obstruction.
   * Inclusion is permitted immediately after unsuccessful attempts at percutaneous recanalization of total occlusions of infra-inguinal arteries.
8. Coagulopathy:

   * aPTT greater than 1.4 x mean laboratory normal reference range
   * International Normalized Ration of Prothrombin Time greater than 1.5
   * Patients on anticoagulation therapy are eligible to participate, with reversal of coagulopathy in accordance with ACC/AHA guidelines, except patients with: Recent arterial (0-1 month) thromboemboism; Recent venous (0-3 months) thromboembolism; Recurrent venous thromboembolism; Non-valvular atrial fibrillation and previous thromboembolism; Mechanical prosthetic valve.
9. Women of childbearing potential.
10. Subjects unwilling to use barrier contraception during the study.
11. Subjects unsuitable for unilateral investigational thigh compression for perfusion measurements due to:

    * Patent femoropopliteal or femorotibial bypass graft or patent femoropopliteal stent on both limbs.
    * Subjects with one of the above features who are amenable to contralateral thigh compression are eligible for enrollment.
12. Immune compromise including chronic HIV, HBV, and HCV infection.
13. Contraindication to Magnetic Resonance Imaging:

    * Allergy to Gadolinium MRI contrast agents.
    * Implanted cardiac pacemaker or defibrillator.
    * Central nervous system aneurysm clips.
    * Implanted neural stimulator.
    * Cochlear implant.
    * Ocular foreign body (e.g. metal shavings).
    * Insulin Pump.
    * Metal shrapnel or bullet.
    * Note: When subjects can provide evidence that their implanted device is labeled compatible with MRI, exceptions to the above exclusions can be made and recorded in the note.
14. Creatinine clearance less than or equal to 20 mL per minute. Creatinine clearance (CLcr) will be estimated using the Cockcroft-Gault formula.
15. Current alcohol, drug abuse, severe medical, psychiatric, behavioral, or emotional disorder of any other condition that may preclude a subject from complying with all requirement of the protocol.
16. Subjects receiving experimental medication or participating in another study receiving an experimental drug or procedure within 30 days prior to enrollment.
17. Unable or unwilling to provide written informed consent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2004-03-27; Study Completion 2011-12-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Baptist Health System, Inc., Birmingham, Alabama
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Background] Anderson WF. What about those monkeys that got T-cell lymphoma? Hum Gene Ther. 1993 Feb;4(1):1-2. doi: 10.1089/hum.1993.4.1-1. No abstract available. PMID 8461379
- [Background] 2nd Euregenethy Multidisciplinary Forum on Regulatory and Safety Issues in Gene Therapy. June 9-11, 2000. Paris, France. Abstracts. J Gene Med. 2000;2(4 Suppl):1-47. No abstract available. PMID 10979487
- [Background] Adam E, Nasz I. [Adenovirus vectors and their clinical application in gene therapy]. Orv Hetil. 2001 Sep 23;142(38):2061-70. Hungarian. PMID 11697063